CLINICAL TRIAL: NCT06874101
Title: Evaluating a Respiratory Oxygen Adherence Monitor for COPD Patients With Long-term Oxygen Therapy
Brief Title: Respiratory Oxygen Adherence Monitor for Chronic Obstructive Pulmonary Disease Patients
Acronym: ROAM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Barron Associates, Inc. (Industry)
Collaborators: University of Virginia (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ROAM; 5R44HL147667-03 (NIH)
Record Dates: First submitted 2025-02-26; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: COPD; COPD - Chronic Obstructive Pulmonary Disease
Keywords: oxygen therapy; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ROAM Group (Experimental): The ROAM group participants will have access to the ROAM user feedback display on their concentrator and portable tank oxygen delivery systems, throughout the 4-week study duration.
  Interventions: Device: Activated ROAM System with User Feedback
- Control Group (Sham Comparator): The control group participants will have their oxygen delivery concentrators and portable tanks fitted with the ROAM system, which will monitor their usage, but they will not receive any of the user feedback or have access to the ROAM software.
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Activated ROAM System with User Feedback — The activated ROAM device will provide the user with daily information about their oxygen therapy usage and pulse oximetry.
  Arms: ROAM Group
Device: Sham Comparator — The sham comparator is a ROAM device that monitors oxygen usage, but keeps the usage details blind to the user.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to test a device called "ROAM" that is being developed to see how patients with chronic obstructive pulmonary disease (COPD) use oxygen therapy over a long period of time. This study will focus on evaluating the ROAM device, which will be attached to your oxygen source. The question that the study aims to answer is: will patients who receive daily adherence feedback from the ROAM have increased adherence to their prescribed long term oxygen therapy regimens?

Researchers will compare the amount of time using oxygen and attitudes about oxygen therapy observed in a group that receives feedback from ROAM, and a control group that does not receive feedback.

Participants will have their oxygen supplies fitted with the ROAM device and then use their oxygen as usual for the 5-week study duration. Participants in the study group will have access to information about their oxygen usage and pulse oximetry levels. All participants will attend two in-clinic sessions of about an hour each, and will complete questionnaires at the beginning and end of the study.

DETAILED DESCRIPTION:
This clinical trial will be a conventional randomized, parallel controlled trial to evaluate the primary hypothesis that a 4-week period of using the ROAM adherence monitor and support system will result in increased adherence when compared to a control group with no adherence monitoring. The participant population will be individuals with chronic obstructive pulmonary disease (COPD), and who have been prescribed oxygen therapy for a minimum of 8 hours/day. Half of the participants will be randomly assigned to the ROAM group; the other half will comprise the control group.

All participants will bring their regular oxygen supplies to the clinic to be fitted with the ROAM sensors. To establish baseline adherence, for the first week, all participants will be blinded to feedback from the ROAM system (including oxygen usage times and oxygen saturation levels); a special code will disable feedback on the local system, including the adherence displays and notifications. After one week, the oxygen usage times will be averaged, and used as a baseline of adherence.

Control participants will continue to be blinded to the ROAM feedback for the next four weeks. After the first week, the ROAM group participants will be instructed to enter a code to enable the ROAM user feedback display on the concentrator and portable tank systems. These participants will be instructed to take pulse oximetry readings as they usually do using the ROAM system's included oximeter. A minimum of two readings per day will be encouraged by built-in alerts on the system. They will continue using the system, while receiving feedback on daily adherence rates and oxygen saturation levels, for the 4-week study duration.

The average daily oxygen use times over the four-week study period will be computed, and use times for the ROAM group will be compared to those of the control group. At the beginning and end of the study, patients will complete a questionnaire to assess attitudes toward treatment. The primary outcome metric will be adherence rates (% adherent = actual treatment time/prescribed treatment time) of the oxygen therapy. The secondary outcome metric will be attitude towards treatment, as assessed via questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Post-Bronchodilator FEV1/FVC<.80
* Participants with medical history of COPD
* Prescription for oxygen use via nasal cannula or mask at home
* At baseline of health with no hospitalization/exacerbation within the past 6 weeks
* Use of Continuous oxygen at baseline

Exclusion Criteria:

* Post -Bronchodilator FEV1/FVC ≤25%
* Intermittent oxygen use at home
* Inability to understand simple instructions
* Respiratory exacerbation or infections within 6 weeks prior to screen visit
* Not at baseline of medical health prior to screen visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adherence rates of oxygen therapy | From enrollment through completion of the study at 5 weeks
  Adherence rates are computed as the participant's average daily actual treatment time divided by the prescribed daily treatment time.

SECONDARY OUTCOMES:
Patient Activation Model Scores | at the study completion at 5 weeks
  The Patient Activation Model (PAM) is an established, highly reliable, questionnaire that reflects a developmental model of patient engagement with their healthcare regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Krepkovich, MS, Principal Investigator — Barron Associates
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No